CLINICAL TRIAL: NCT05069077
Title: the Effect of Music on Pain and Women Satisfaction During Diagnostic Outpatient Hysteroscopy in Postmenopausal Women: a Randomized Controlled Trial
Brief Title: the Effect of Music on Pain and Women Satisfaction During Diagnostic Outpatient Hysteroscopy in Postmenopausal Women
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: consensus between researchers. Limited time and resources
Sponsor: Cairo University (Other)
Collaborators: Hospital El Gezeera (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, assistant professor of obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: hysteroscopy menopause 8233
Record Dates: First submitted 2021-09-25; First posted 2021-10-06 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Hysteroscopy
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- music group (Experimental): In the music group, music chosen by the participant will be played through a speaker by the nursing staff during outpatient hysteroscopy. Music will be played through a speaker instead of headphones in order to maintain good communication and interaction between the participant and the doctor.
  Interventions: Other: Music
- non-music group (Other): Participants in the non-music group will undergo diagnostic outpatient hysteroscopy in the same setting and standard procedure without listening to any music.
  Interventions: Other: No music

INTERVENTIONS:
Other: Music — In the music group, music that chosen by the participant will be played through a speaker by the nursing staff during outpatient hysteroscopy. Music will be played through a speaker instead of headphones in order to maintain good communication and interaction between the participant and the doctor.
  Arms: music group
Other: No music — Participants in the non-music group will undergo outpatient hysteroscopy in the same setting and standard procedure without listening to any music.
  Arms: non-music group

SUMMARY:
The aim of this study is to demonstrate the value of music in diagnostic outpatient hysteroscopy on patients' level of pain and satisfaction in postmenopausal women

ELIGIBILITY:
Inclusion Criteria:

* Menopausal patients with an indication for ofﬁce hysteroscopy (postmenopausal bleeding or abnormal ultrasound ﬁndings)

Exclusion Criteria:

* patients with cervical pathology retroverted uterus (detected by transvaginal ultrasound) previous cervical surgery patients with severe vaginal bleeding

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-15 (Estimated); Primary Completion 2022-05-10 (Estimated); Study Completion 2022-05-15 (Estimated)

PRIMARY OUTCOMES:
Intensity of pain | 5 minutes
  Pain intensity will be assessed by visual analog scale during the procedure. visual analog scale ranging from 0 to 100

SECONDARY OUTCOMES:
Intensity of pain | 20 minutes
  Pain intensity will be assessed by visual analogue scale during the procedure.visual analogue scale ranging from 0 to 100